CLINICAL TRIAL: NCT03301194
Title: In-depth Study of the Cost-effectiveness of the Risk Assessment and Management Programme for Hypertension (RAMP-HT) for Patients With Uncontrolled Hypertension in Primary Care in Hong Kong
Brief Title: Cost-effectiveness of RAMP-HT for Patients With Uncontrolled Hypertension in Hong Kong
Status: Completed | Type: Observational
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. YU Yee Yak, Esther, Clinical Assistant Professor, The University of Hong Kong
Other Study IDs: HKUCTR-2233
Record Dates: First submitted 2017-09-27; First posted 2017-10-04 (Actual); Last update posted 2019-05-03 (Actual); Status verified 2019-05

CONDITIONS: Hypertension; Cost Effectiveness
Keywords: Hypertension; Effectiveness; Cost Effectiveness; Cost; Multi-disciplinary; Risk Stratification
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- RAMP-HT patients: HT patients who have enrolled into the RAMP-HT between 1 October 2011 and 31 March 2012 and fulfilled the inclusion criteria and without any exclusion criteria
  Interventions: Other: RAMP-HT
- Usual care patients: HT patients receiving usual care in GOPCs who have never enrolled into RAMP-HT on or before 31 March 2017 and fulfilled the inclusion criteria and without any exclusion criteria

INTERVENTIONS:
Other: RAMP-HT — RAMP-HT was launched since October 2011 by the Hospital Authority with the support from the Food and Health Bureau. Standardized cardiovascular risk factor assessment, hypertensive complication screening and assessment on patient adherence to treatment are carried out on enrolled patients. Patients are stratified into low, medium or high risk groups according to the 10-year cardiovascular disease (CVD) risk calculated from their relevant risk factors by the Joint British Society 2005 Equation. A multidisciplinary team comprised of doctors, nurses, dieticians, physiotherapists and/or occupational therapists would then deliver individualized management targeted to the patient's risk factors according to standardized risk-stratified guidelines.
  Groups: RAMP-HT patients

SUMMARY:
Hypertension (HT) is an important risk factor for stroke, coronary heart disease (CHD), heart failure and renal diseases, and the leading risk factor of global disease burden. A multitude of interventions have proven efficacy in lowering blood pressure and reducing long term HT complications, including pharmacologic treatment, DASH diet (Dietary Approaches to Stop Hypertension), exercise, weight reduction, smoking cessation, alcohol moderation and self-monitoring of blood pressure.

Objectives:

To evaluate long-term effectiveness and cost-effectiveness of Risk-Assessment-and-Management-Programme-for-Hypertension (RAMP-HT), a multi-disciplinary structured service to enhance quality of hypertension care in primary care compared to usual care

Hypotheses:

1. RAMP-HT is effective in reducing HT complications, based on previous results showing RAMP-HT was effective in improving patients' blood pressure
2. RAMP-HT is cost-effective

Design and Subjects:

Retrospective study of 5-year longitudinal data on matched cohorts of public primary care patients with uncontrolled HT under RAMP-HT and usual care will be conducted to evaluate long-term effectiveness and direct medical costs. Results from the long-term effectiveness and costing analyses will be applied to Markov modeling to determine the life time cost-effectiveness of RAMP-HT.

Main outcome measures:

1. 5-year incidence of cardiovascular complications
2. Direct medical costs of RAMP-HT and usual care HT patients
3. Incremental cost-effectiveness ratio (ICER) of cost per quality-adjusted life year (QALY) gained by RAMP-HT compared to usual care

Data analysis:

Cox regression will be performed to estimate the effect of RAMP-HT on the development of HT complication adjusted for baseline covariates. Descriptive statistics will be used to calculate costs of RAMP-HT and annual direct medical costs for HT patients. Markov modeling will be used to simulate 2 patient cohorts (RAMP-HT versus usual care) to estimate the respective lifetime direct medical costs and QALY gained/person. Cost/QALY of RAMP-HT will be compared to that of usual care to determine the ICER.

Expected results:

The results can provide evidence on the effectiveness and cost-effectiveness of RAMP-HT for primary care patients with uncontrolled HT, which can inform health policy and service planning.

DETAILED DESCRIPTION:
Aim and objectives:

The aim of this study is to evaluate the cost-effectiveness of the RAMP-HT of the HA in primary care patients with uncontrolled hypertension.

The objectives are to:

1. Evaluate the long term (5-year) effectiveness of RAMP-HT compared to usual care in reducing cardiovascular complications, end-stage renal disease and all-cause mortalities in a cohort of primary care patients with uncontrolled hypertension at baseline
2. Estimate the direct medical cost of RAMP-HT and other health services among primary care HT patients with or without complications
3. Evaluate the cost-effectiveness of RAMP-HT, compared to usual care, in gaining one QALY in primary care patients with uncontrolled hypertension

Hypotheses:

1. RAMP-HT is more effective in reducing 5-year cardiovascular complications, end stage renal disease and all-cause mortality among primary care patients with uncontrolled hypertension compared to usual care
2. The direct medical cost of RAMP-HT patients, for the same disease complication status, is not higher than that of usual care except for the RAMP-HT cost
3. The direct medical cost of HT patients with one or more complications is higher than that of HT patients without any complication
4. RAMP-HT is cost-effective compared to usual care, i.e. ICER per QALY gained is below the threshold value of 1 annual GDP (Gross Domestic Product) per capita of Hong Kong, which is the benchmark recommended by the World Health Organization

ELIGIBILITY:
Inclusion criteria:

1. Age ≥ 18 years old and < 80 years old
2. Coded with ICPC-2 of K86 on or before baseline*
3. Had uncontrolled blood pressure (i.e. average Systolic Blood Pressure (SBP) ≥ 140mmHg OR Diastolic Blood Pressure (DBP) ≥ 90mmHg between 6 months before and 3 months after baseline*)

Exclusion criteria:

1. Patients who had a diagnosis of any HT complications defined by relevant ICPC-2 and/or ICD-9-CM diagnosis codes on or before baseline*
2. Patients diagnosed to have Diabetes Mellitus (DM) on or before 31 March 2017, defined by ICPC-2 codes of T89 or T90
3. Patients exclusively managed by Specialist Out-Patient Clinic (SOPC) on or before baseline*

   * Baseline: date of RAMP-HT enrolment for RAMP-HT cohort, and 31 March 2012 for usual care cohort

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients who have enrolled into the RAMP-HT between 1 October 2011 and 31 March 2012, fulfilled the inclusion criteria and without any exclusion criterion will be included in the RAMP-HT cohort. The same number of matched patients receiving usual care in general outpatient clinics (GOPCs) who have never enrolled into RAMP-HT on or before 31 March 2017, fulfilled the inclusion criteria and without any exclusion criterion will be randomly selected from the HA clinical management system (CMS) to form the usual care cohort.
Sampling Method: Probability Sample
Enrollment: 158322 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
The 5-year incidence of CVD among RAMP-HT and usual care HT patients | 60-month
  CVD is defined as the presence of any of coronary heart disease (CHD), heart failure or stroke. CHD includes all ischaemic heart disease, myocardial infarction, coronary death or sudden death as indicated by the ICPC-2 K74 to K76 or ICD-9-CM 410.x, 411.x to 414.x, 798.x codes. Heart failure is defined as the ICPC-2 K77 or ICD-9-CM 428.x codes. Stroke (fatal and non-fatal stroke) is defined by the ICPC-2 K89 to K91 or ICD-9-CM 430.x to 438.x codes.
The direct medical costs of RAMP-HT and usual care HT patients with and without complications | 12-month before baseline, baseline, 12, 24, 36, 48 and 60-month
  Public medical costs will be estimated from products of the unit costs (published in the HKSAR Government Gazette and Hospital Authority (HA) ordinance (Chapter 113) of charges for non-entitled persons) and the utilization rates of 1) dispensed drugs, 2) laboratory tests and investigations, 3) healthcare services including general outpatient clinics (GOPC), specialist outpatient clinics (SOPC), allied health services (e.g. dietician, physiotherapist or occupational therapist), accident and emergency (A&E) department and 4) admissions to hospital in the 12 months before baseline and at 12, 24, 36, 48 and 60 months after study enrolment for each patient in the study cohorts.
  Private direct medical costs include the cost of all private Western doctor and Chinese medicine practitioner consultations, private hospitalisation and self-medications inclusive of self-financed medications prescribed by the HA.
The ICER of cost per QALY gained by RAMP-HT compared to usual care group | 60-month
  The ICER was the ratio of the incremental costs of RAMP-HT group over the incremental effectiveness compared to those of the usual care group. In this study, the ICER referred to 1) program cost per HT-related complication reduced by RAMP-HT, and 2) program cost per event-free year in the RAMP-HT group, compared to the usual care group.

SECONDARY OUTCOMES:
The 5-year incidence of end stage renal disease (ESRD) and all-cause mortality among RAMP-HT and usual care HT patients | 60-month
  ESRD is defined by any of ICD-9-CM 250.3x, 585.x, 586.x, or an estimated Glomerular Filtration Rate (eGFR) < 15mL/min/1.73m2, according to the definition of the National Kidney Foundation. Mortality is defined by a documented death in the Hong Kong Death Registry.
The hazard ratio of CVD, ESRD and all-cause mortalities between RAMP-HT and usual care group | 60-month
  Multivariable Cox proportional hazards regression will be performed to estimate the adjusted effect of RAMP-HT on the dependent variable of each first HT complication event, adjusting for all baseline covariates of patients.
The Number-Need-to-Treat (NNT) to reduce one CVD, ESRD and mortality in 5 years by RAMP-HT | 60-month
  NNT is the average number of patients who need to be treated to prevent one additional outcome event. It is defined as the inverse of the absolute risk reduction.

CONTACTS AND LOCATIONS:
Overall Officials: Esther Yee Tak Yu, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-03-04): https://cdn.clinicaltrials.gov/large-docs/94/NCT03301194/Prot_SAP_000.pdf